CLINICAL TRIAL: NCT04857606
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 609 in Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: Single Ascending Dose of AMG 609 in Participants With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20200001
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Single ascending dose; NAFLD; AMG 609
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMG 609 (Experimental): Up to 7 cohorts ranging by various dose levels.
  Interventions: Drug: AMG 609
- Placebo (Experimental): Participants will receive the matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 609 — Single dose of AMG 609 administered as a subcutaneous injection.
  Arms: AMG 609
Drug: Placebo — Single dose of placebo administered as a subcutaneous injection.
  Arms: Placebo

SUMMARY:
This study aims to assess the safety and tolerability of AMG 609 when administered subcutaneously as single doses in participants with non-alcoholic fatty liver disease (NAFLD).

ELIGIBILITY:
* Inclusion Criteria

  * Men and women age ≥ 18 to ≤ 70 years of age at the time of signing the informed consent
  * Body mass index (BMI) of ≥ 27 kg/m2 to ≤ 45.0 kg/m2
  * Liver steatosis, measured by MRI-PDFF, greater than 8%
* Exclusion Criteria

  * Evidence of other liver disease (eg, viral hepatitis, primary sclerosing cholangitis, primary biliary cholangitis, autoimmune chronic hepatitis, Wilson's disease, alpha-1 anti-trypsin deficiency, haemochromatosis, drug-induced liver injury, bile duct obstruction, known or suspected hepatocellular carcinoma).
  * Significantly elevated LFTs (more than 1.5x ULN)
  * Uncontrolled diabetes (HgbA1c > 9%) or uncontrolled hypertension.
  * History of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers occurring more than 5 years prior to randomization or 3 years prior to randomization for basal cell carcinoma.
  * Females of reproductive potential.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Subject Incidence of Treatment-emergent Adverse Events | Day 1 to Day 150
Subject Incidence of Clinically Significant Change from Baseline in Laboratory Analytes | Baseline to Day 150
Subject Incidence of Clinically Significant Change from Baseline in Vital Signs | Baseline to Day 150
Subject Incidence of Clinically Significant Change from Baseline in 12-lead Electrocardiograms (ECGs) | Baseline to Day 113

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of AMG 609 | Up to Day 150
Time to Maximum Observed Concentration (Tmax) of AMG 609 | Up to Day 150
Area Under the Concentration Time Curve (AUC) of AMG 609 | Up to Day 150

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (10):
  - The Institute for Liver Health - Arizona Liver Health, Chandler, Arizona
  - ProSciento Incorporated, Chula Vista, California
  - Catalina Research Institute, Montclair, California
  - Inland Empire Liver Foundation, Rialto, California
  - Orange County Research Center, Tustin, California
  - Translational Clinical Research LLC, Aventura, Florida
  - Texas Liver Institute, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - McGuire VA Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com